CLINICAL TRIAL: NCT05121415
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: Investigation of Genetic Disease Marker Associated With Spontaneous Haemorrhagic Stroke Complicating Severe Pre-eclampsia in Pregnancy
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1189
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Hemorrhagic Stroke; Eclampsia
Keywords: SNP
MeSH Terms: conditions — Hemorrhagic Stroke; Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: patients with hemorrhagic stroke complicating severe pre-eclampsia in pregnancy
  Interventions: Genetic: SNP analysis of the DNA
- Control group: patients without hemorrhagic stroke complicating severe pre-eclampsia in pregnancy
  Interventions: Genetic: SNP analysis of the DNA

INTERVENTIONS:
Genetic: SNP analysis of the DNA — SNP analysis of the DNA obtained from peripheral blood sample

SUMMARY:
To search for a genetic marker of hemorrhagic stroke complicating severe eclampsia, a single nucleotide polymorphism (SNP) analysis of DNA obtained from the peripheral blood of patients with hemorrhagic stroke and normal control will be performed.

DETAILED DESCRIPTION:
Detailed Description:

Unrelated Korean subjects who have Spontaneous hemorrhagic stroke complicating severe eclampsia in pregnancy were recruited in the current study. Genotyping for various SNP associated due to the linkage disequilibrium patterns is to be performed. Genotypes would be statistically compared between patients with hemorrhagic stroke and normal control subjects free of hemorrhagic stroke

ELIGIBILITY:
Inclusion Criteria:

-patients with hemorrhagic stroke complicating severe eclampsia in pregnancy

Exclusion Criteria:

patients without hemorrhagic stroke complicating severe eclampsia in pregnancy

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: patients with hemorrhagic stroke complicating severe eclampsia in pregnancy who visited Scientific Center for Obstetrics, Gynecology and Perinatology. Kazakhstan, Almaty
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
genotyping for the SNP associated with hemorrhagic stroke complicating severe eclampsia in pregnancy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aygul Terlikbayeva, PhD, Study Director — JSC "Scientific center of obstetrics, gynecology and perinatology"
Locations (1):
- Hospital, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided